CLINICAL TRIAL: NCT01006655
Title: The Effect of HFA - Beclomethasone Dipropionate - Qvar - on Bronchial Hyperreactivity in Preschool Children
Brief Title: The Effect of HFA - Beclomethasone Dipropionate Qvar on Bronchial Hyperreactivity in Preschool Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, l_bentur, Head of pediatric pulmonary institute, Ruth children hospital, Rambam Health Care Campus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: qvar-adenosineCTIL
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Asthma; Bronchial Hyperresponsiveness
Keywords: asthma; preschool children; bronchial hyperresponsiveness; beclometasone dipropionate - HFA; Qvar; Adenosine Challenge test
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo, adenosine challenge test (Placebo Comparator): Controlled or partially controlled multiple trigger wheezing children received 4 weeks of placebo, preceded and succeeded by AMP challenge test,
  Interventions: Drug: placebo
- Qvar, adenosine challenge test (Active Comparator): Patients will receive 4 weeks of inhale QVAR (HFA beclomethasone) 100µg through a spacer device, twice a day
  Interventions: Drug: Beclomethasone dipropionate HFA

INTERVENTIONS:
Drug: Beclomethasone dipropionate HFA — 100µg twice a day, through inhaler autohaler, using a spacer device, preceded and followed by adenosine challenge test
  Other Names: Qvar
  Arms: Qvar, adenosine challenge test
Drug: placebo — inhalation twice a day for one month, preceded and followed by adenosine challenge test
  Arms: placebo, adenosine challenge test

SUMMARY:
Respiratory diseases including Asthma are high prevalent among preschool children. Specific treatment, nowadays, include steroid inhalers and anti leukotrienes. It is known that the amount of the drug reaching small airways and lungs is bigger how much smaller the particles liberated by inhalers. Beclometasone is being used for treating asthma for 30 years. Lately emerged a new presentation of beclometasone, which liberates particles as small as 2.1 µg, that is supposed to reach the small airways at higher concentrations and be more suitable to patients who don't cooperate properly to the procedure of inhalation.

The investigators' group has reported successfully the possibility to perform Pulmonary Challenge tests (adenosine, methacholine and exercise) in tender age. Other studies reported relation between asthma control and reduction in airway hyperreactivity. The purpose of this study is to evaluate the efficacy of Beclometasone dipropionate - Qvar to reduce airways hyperreactivity in preschool children, as demonstrated by adenosine challenge test.

DETAILED DESCRIPTION:
26 - 30 patients, between 3 -6 years old, mild asthmatics, with positive adenosine challenge test, will received in a randomized, double blind, cross over assignment Beclometasone dipropionate (100µg twice a day) or placebo, through an inhaler (autohaler) device, attached to a spacer device, during four consecutive weeks. Adenosine Challenge test will be performed another time at the end of this four weeks period. After 2 weeks with no medication (wash out period) the patients will receive the second intervention (beclometasone dipropionate or placebo) in a cross over manner and will be submitted to the last adenosine challenge test.

Clinical evaluation, resting spirometry and subjective evaluation through an analogical symptoms scale will be recorded in each visit.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of mild asthma
* children aged between 3 - 6 years old
* able to perform spirometry and adenosine challenge test
* positive challenge test at the time of inclusion
* without prophylactic treatment for asthma
* signed informed consent to join the research by the parents or legal tutor

Exclusion Criteria:

* other chronic diseases
* use of oral steroids in the last two months
* emergency room visit in the last two months
* pneumonia in the last two months
* impossibility to perform lung function tests
* disagreement of the parents or legal tutor

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Background] Menzies D, Nair A, Hopkinson P, McFarlane L, Lipworth BJ. Differential anti-inflammatory effects of large and small particle size inhaled corticosteroids in asthma. Allergy. 2007 Jun;62(6):661-7. doi: 10.1111/j.1398-9995.2007.01376.x. PMID 17508971
- [Background] Koh YY, Lee MH, Sun YH, Park Y, Kim CK. Improvement in bronchial hyperresponsiveness with inhaled corticosteroids in children with asthma: importance of family history of bronchial hyperresponsiveness. Am J Respir Crit Care Med. 2002 Aug 1;166(3):340-5. doi: 10.1164/rccm.2101158. PMID 12153967
- [Background] Hakim F, Vilozni D, Adler A, Livnat G, Tal A, Bentur L. The effect of montelukast on bronchial hyperreactivity in preschool children. Chest. 2007 Jan;131(1):180-6. doi: 10.1378/chest.06-1402. PMID 17218573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from Pediatric pulmonology out clinic, Rambam Medical Center, Haifa, Israel between March 2009 and January 2010
Pre-assignment Details: 40 participants approached, 23 agreed and have been screened, 2 excluded (1 adenosine challenge test negative, 1 obstructive respiratory impairment)
Groups:
- Placebo First, Adenosine Challenge Test: 11 controlled or partially controlled multiple trigger wheezing children received 4 weeks of placebo, preceeded and succeeded by AMP challenge test, followed by an equal period of QVAR and another AMP challenge test
- Qvar First, Adenosine Challenge Test: 10 controlled or partially controlled multiple trigger wheezing children received 4 weeks of QVAR, preceeded and succeeded by AMP challenge test, followed by an equal period of Placebo and another AMP challenge test
Period: First Intervention
Arm/Group | Placebo First, Adenosine Challenge Test | Qvar First, Adenosine Challenge Test
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Placebo First, Adenosine Challenge Test | Qvar First, Adenosine Challenge Test
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Adenosine Challenge Test | Qvar First, Adenosine Challenge Test
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First, Adenosine Challenge Test | Qvar First, Adenosine Challenge Test | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 10 | 21
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.94 (1.08) | 5.05 (1.05) | 4.95 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  Israel | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Adenosine Challenge Test
Description: Adenosine challenge test were measured and described as PC 20 - the concentration that corresponded to a FEV1 impairment equal or bigger than 20%. The stage was also recorded
Time Frame: ten weeks
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Placebo First, Adenosine Challenge Test | Qvar First, Adenosine Challenge Test
Number analyzed (Participants) | 11 | 11
mg/ml | 18.46 (26.17) | 142.61 (71.6)

ADVERSE EVENTS:
Arm/Group | Placebo First, Adenosine Challenge Test | Qvar First, Adenosine Challenge Test
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No